CLINICAL TRIAL: NCT01234506
Title: Community Alliance for Quality of Life in Long Term Care: Oxidative Stress and Nutritional Supplementation Intervention Study
Brief Title: Oxidative Stress and Nutritional Supplementation Intervention Study
Acronym: Oxi-Stress
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other)
Responsible Party: Principal Investigator, Susan Whiting, PhD, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NHPD-150212
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Oxidative Stress; Inflammation; Aging; Dementia; Pain
Keywords: long term care; lignans; oxidative stress; inflammation; aging; dementia; postural balance; depression; muscle weakness; quality of life; pain
MeSH Terms: conditions — Inflammation; Dementia; Pain; Depression; Muscle Weakness | interventions — secoisolariciresinol diglucoside

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- secoisolariciresinol diglucoside (Active Comparator): Secoisolariciresinol diglucoside (SDG) supplementation as 0.8g/day of BeneFlax containing 300 mg SDG. 1000 IU vitamin D as standard of care.
  Interventions: Dietary Supplement: secoisolariciresinol diglucoside
- Placebo (Placebo Comparator): An equal volume of measured whey protein (unflavored) to the Beneflax and 1000 IU vitamin D as standard of care.
  Interventions: Dietary Supplement: secoisolariciresinol diglucoside

INTERVENTIONS:
Dietary Supplement: secoisolariciresinol diglucoside — SDG supplementation as a packet of 0.8g/day of BeneFlax containing 300 mg SDG for 24 weeks
  Other Names: Beneflax Flax Lignan Extract Archer Daniels Midland,#080001.; Natural Factors Whey Factors whey protein (unflavored).; Vitamin D NPN 80003663 WN Pharmaceuticals

SUMMARY:
A major means whereby oxidative stress promotes aging-related disease is by activating inflammatory pathways. Decreasing oxidative stress and inflammation should ameliorate many of the problems associated with aging, including vascular dementia, Alzheimer's disease, osteoporosis, muscle wasting, insulin resistance, type 2 diabetes, and metabolic syndrome. Animal and human studies have demonstrated that consumption of vitamin D and phase 2 protein inducers decrease oxidative stress and associated inflammation. The flax lignan secoisolariciresinol diglucoside (SDG) is metabolized to enterolactone, a potent phase 2 protein inducer. Animal and human studies have shown that consumption of flax seed or its component SDG decreases hypertension, serum cholesterol, atherosclerosis, the growth of experimentally-induced cancers as well as metastases of human breast tumours implanted into nude mice, and delays the development of type 2 diabetes. Vitamin D plays a role in modulating inflammation, enhancing immunity (while suppressing autoimmune injury) and exerting control over cell differentiation. Adequate levels of vitamin D also appear to promote better glycemic control. The investigators predict that consumption of SDG in persons with adequate vitamin D status will decrease oxidative stress and associated inflammation. If this hypothesis is upheld, this research has the potential to greatly decrease healthcare costs while allowing healthier aging.

ELIGIBILITY:
Inclusion Criteria:

* adults residing in a long term care facility
* resident for a minimum of four weeks prior to entry
* able to comply with study protocol
* able to follow simple instructions
* able to give informed consent or has a legally acceptable representative who is able to provide consent

Exclusion Criteria:

* Age below 60 or above 80 years.
* Individuals at risk of hypotension or with symptomatic hypotension.
* Fasting hypoglycemia.
* Unstable diabetes
* Diabetics taking insulin
* Current cancer or diagnosed with cancer in the past 2 years.
* Women with an immediate family history or personal history of breast cancer or ovarian cancer
* Significant liver disorder
* Significant gastrointestinal disorder including inflammatory bowel disease but not constipation
* Significant kidney disorder
* Unstable or severe cardiac disease, recent MI or stroke either in past 6 months or significantly (i.e., severely) affecting physical mobility.
* Unstable other medical disease including, but not limited to, pulmonary disorder, epilepsy and genitourinary disorder.
* Migraine with aura within the last year (as this is a risk factor for stroke).
* Current diagnosis of a bleeding condition, or at risk of bleeding.
* Significant immunocompromise.
* Other unstable conditions.
* Current use of hormone replacement therapy except thyroid medication
* Current use of warfarin, clopidogrel, ticlopidine, dipyridamole or their analogues.
* Intolerances or allergies to flax or vitamin D.
* Estimated probability of longevity of less than one year based on medical opinion

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety of consumption of 300 mg/day of the flax lignan secoisolariciresinol diglucoside (SDG) in older adults (60-80 y) | 24 weeks
  Adverse event occurrences will be compared descriptively between the SDG and placebo groups. Safety will be assessed at 0, 6, 12, 18 and 24 weeks; as part of the blood collection (urea, creatinine, total bilirubin, platelets, hematocrit, haemoglobin, mean corpuscular haemoglobin, mean corpuscular volume, white blood cell count, total protein including albumin and prealbumin, total calcium, electrolytes, glucose, liver enzymes (AST, ALT, ALP), total protein, albumin, lipids, HbA1c (for diabetic participants). Blood pressure measurements will be performed every two weeks
Effect of SDG on oxidative stress and inflammation | 24 weeks
  SDG and placebo groups will be compared at 0, 12 and 24 weeks for changes in oxidative stress measurements (plasma malondialdehyde), pro-inflammatory markers (IL-6, IL-1α, IL-1β, 8-isoprostane, TNF-α, C-reactive protein).

SECONDARY OUTCOMES:
Effect of SDG on quality of life | 24 weeks
  SDG and placebo groups will be compared at 0, 12 and 24 weeks for changes in cognitive function, pain, and physical function including falls, as well as performance of activities of daily living.
Effect of SDG supplement on blood levels of flax lignan metabolites | 24 weeks
  To further understand the pharmacology of SDG, we will analyze plasma levels of the SDG metabolites secoisolariciresinol, enterolactone and enterodiol in those subjects given flax lignan supplement. Levels will be determined 0, 12 and 24 weeks.
To measure effects of SDG on bone resorption | 24 weeks
  SDG and placebo groups will be compared at 0 and 24 weeks for changes in bone resorption as assessed by measurement of cross-linked N-telopeptides type I collagen serum levels.
Effect of SDG on blood lipids | 24 weeks
  SDG and placebo groups will be compared at 0, 12 and 24 weeks for changes in nonfasting levels of cholesterol, LDL, HDL, and triglycerides.

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Whiting, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- Saskatoon Health Region, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Adolphe JL, Whiting SJ, Juurlink BH, Thorpe LU, Alcorn J. Health effects with consumption of the flax lignan secoisolariciresinol diglucoside. Br J Nutr. 2010 Apr;103(7):929-38. doi: 10.1017/S0007114509992753. Epub 2009 Dec 15. PMID 20003621
- [Result] Di Y, Jones J, Mansell K, Whiting S, Fowler S, Thorpe L, Billinsky J, Viveky N, Cheng PC, Almousa A, Hadjistavropoulos T, Alcorn J. Influence of Flaxseed Lignan Supplementation to Older Adults on Biochemical and Functional Outcome Measures of Inflammation. J Am Coll Nutr. 2017 Nov-Dec;36(8):646-653. doi: 10.1080/07315724.2017.1342213. Epub 2017 Sep 18. PMID 28922068
- [Result] Alcorn J, Whiting S, Viveky N, Di Y, Mansell K, Fowler S, Thorpe L, Almousa A, Cheng PC, Jones J, Billinsky J, Hadjistavropoulos T. Protocol for a 24-Week Randomized Controlled Study of Once-Daily Oral Dose of Flax Lignan to Healthy Older Adults. JMIR Res Protoc. 2017 Feb 3;6(2):e14. doi: 10.2196/resprot.6817. PMID 28159728